CLINICAL TRIAL: NCT02498366
Title: Exertional Rhabdomyolysis- Characterization of Prediction Tests for Return to Duty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2388-15-SMC
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental protocol (Experimental): 50 healthy, male, trained and aged 18-30 will be recruited and asked to undergo a series of physical tests.
  Interventions: Other: physical tests

INTERVENTIONS:
Other: physical tests — each subject will undergo the following physical tests: day 1 - anthropometric measurements, wingate test and after 1 hour rest VO2max test. lactic acid levels will be measured before and after both tests.
  day 2 - step test day 3 - running on the anaerobic threshold. blood sample, lactic acid level (measured in blood drop - finger sting) and urine sample will be taken before and after every test in days 2 and 3.

SUMMARY:
In order to determine norm values for skeleton muscle disassembly due to physical exertion in healthy and trained population, and developing a prediction test for approval for rhabdomyolysis injuries to return to duty, 50 healthy subjects will undergo a series of different physical tests.

DETAILED DESCRIPTION:
50 healthy civilians volunteers will be recruited for this study. Each subject will undergo the physical tests: anthropometric measurements, wingate test, VO2max test, step test and running on the anaerobic threshold, on separate days. Blood sample, lactic acid level (measured in blood drop - finger sting) and urine sample will be taken before and after every test.

ELIGIBILITY:
Inclusion Criteria:

* healthy civilians ages 18-30.
* above average aerobic and anaerobic fitness.
* Without heart, cardiovascular, metabolic or respiratory illnesses.
* Without known medical illness or medication use that might endanger the participants.

Exclusion Criteria:

* existence of any of undesired conditions detailed in the inclusion criteria.
* the physician decision.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
creatine phosphokinase (CPK) | 5 experiment days for each subject
  CPK is a marker for muscle damage assessed in blood test. blood sample will be taken before and after step test and running on the anaerobic threshold test.
oxygen consumption (VO2) | 5 experiment days for each subject
  VO2 will be monitored continuously using a metabolic system (ERGOTEST 680, ZAN, GERMANY ) during VO2max test, step test and running on the anaerobic threshold test.

SECONDARY OUTCOMES:
lactic acid | 5 experiment days for each subject
  lactic acid level is assessed from blood drop (finger sting), will be taken before and after every test. lactic acid is a marker for anaerobic effort evaluating.
Myoglobin | 5 experiment days for each subject
  marker from urine sample, taken before and after step test and running on the anaerobic threshold test.
Heart rate | 5 experiment days for each subject
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel